CLINICAL TRIAL: NCT04448392
Title: Evaluation of the Pharmacokinetics and Pharmacodynamics of Valacyclovir in Neonates With Neonatal Herpes Simplex Virus Disease Who Have Completed Standard of Care Treatment With Acyclovir
Brief Title: Valacyclovir in Neonatal Herpes Simplex Virus Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Richard J Whitley, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 300005567; 311653000 (Other: UAB)
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Herpes Simplex Infection
Keywords: valacyclovir
MeSH Terms: interventions — Valacyclovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neonatal HSV disease requiring suppressive therapy (Other): All subjects enrolled in the study will receive 2 (up to 7) days of valacyclovir 20 mg/kg every 8 hours after completion of standard of care treatment course with acyclovir.
  Interventions: Drug: Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir — Upon completion of standard of care acyclovir for treatment of neonatal HSV disease, valacyclovir oral suspension (per ASHP recipe), 20 mg/kg every 8 hours, to be given for 2 (up to 7) days

SUMMARY:
This is an open-label, single center, pharmacokinetic (PK) study to assess valacyclovir pharmacokinetics and pharmacodynamics in neonates and compare to the pharmacokinetics and pharmacodynamics of the standard of care treatment dose of intravenous acyclovir. 6 (up to 10 infants) with virologically confirmed neonatal herpes simplex virus (HSV) disease who meet all inclusion/exclusion criteria will be enrolled in the study. Study duration is 5 years. Primary objective is to define the pharmacokinetics of valacyclovir and assess its safety in neonates 2-12 weeks of age who are ≥ 34 weeks gestation.

DETAILED DESCRIPTION:
This is an open-label, single center, PK study to assess valacyclovir pharmacokinetics and pharmacodynamics in neonates and compare to the pharmacokinetics and pharmacodynamics of the standard of care treatment dose of intravenous acyclovir. Only those babies with virologically confirmed neonatal HSV disease will be enrolled in the study. The decision to initiate valacyclovir for 2 (up to 7) days will be made by a physician based on inclusion/exclusion criteria, and those who meet entry criteria will be eligible for the study. Those enrolled in the study will have daily random parenteral acyclovir PK levels drawn during the first week of treatment (drawn only at times of other lab draws). These infants will also have a pharmacokinetic sampling profile obtained on or after dose 22 and before dose 42 of intravenous acyclovir. The PK samples for the sampling profile will be collected just prior to the next dose of intravenous acyclovir (within 30 minutes prior to the start of the infusion), within 15 minutes of completion of the infusion, and 3-4 hours after infusion. Upon completion of the recommended treatment course duration with intravenous acyclovir determined by disease classification (skin, eye, and mouth; central nervous system; or disseminated disease), the infant will be started on enteral valacyclovir 20 mg/kg every 8 hours.

On day 2 and no more than day 7 of valacyclovir 20 mg/kg every 8 hours, a pharmacokinetic sampling profile will be obtained. The PK samples will be collected just prior to the enteral dose of valacyclovir (hour 0; 8 hours after previous dose and immediately before next dose), 1-2 hours after dose, and 3-5 hours after dose. Primary objective is to define the pharmacokinetics of valacyclovir and assess its safety in neonates 2-12 weeks of age who are ≥ 34 weeks gestation. Secondary objectives are to: 1) assess the pharmacokinetics of high-dose parenteral acyclovir in neonates ≥ 34 weeks gestation with virologically confirmed neonatal HSV disease who are receiving acyclovir as standard of care, 2) compare the pharmacokinetics of high-dose parenteral acyclovir to the pharmacokinetics of the proposed study dose of valacyclovir (20 mg/kg every 8 hours).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parent(s) or legal guardian(s)
* Confirmation of HSV infection from surface culture/PCR, skin lesion culture/PCR, blood PCR, or CSF PCR (performed at UAB Virology lab)
* ≥34 weeks gestational age at birth
* Weight at study enrollment is ≥ 2000 grams
* Receiving intravenous acyclovir, prescribed by the patient's physician for ≤ 14 days
* ≤ 42 days of age at initiation of parenteral acyclovir
* Creatinine ≤ 1.2

Exclusion Criteria:

* Imminent demise
* Current receipt of other investigational drugs
* Major congenital anomaly that in the site investigator's opinion may impact drug metabolism or the patient's volume of distribution
* Creatinine of > 1.2 prior to initiation of valacyclovir
* Evidence of immunosuppression (HIV infected, immune deficiencies, etc.)
* Any condition that, in the opinion of the investigator, would place the subject at an unacceptable injury risk or that may interfere with successful study completion
* > 42 days of age at initiation of parenteral acyclovir
* Concern for parental/guardian compliance

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitley, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama - Children's of Alabama, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
Age, Customized [Count of Participants; unit: Participants] — Age at time of diagnosis of neonatal HSV disease
  Participants
    0-20 days | 4
    21-42 days | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Age at time of parental acyclovir profile (days) [Median (Full Range); unit: days] | 30 [13 to 39]
Age at time of valacyclovir profile (days) [Median (Full Range); unit: days] | 35 [19 to 48]
Interval between parental acyclovir and valacyclovir profile (days) [Mean (Full Range); unit: days] | 6 [3 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve Following Administration of Oral Valacyclovir Suspension 20 mg/kg Every 8 Hours
Description: Blood will be collected to determine the drug concentration of acyclovir, the metabolite of valacyclovir and will include AUC.
Time Frame: Between Day 2 and Day 7 of valacyclovir administration: 0, 1-2, 3-5 hours.
Measure: Mean (Standard Deviation); unit: mgxh/l
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
mgxh/l | 28.8 (16.8)

2. Primary Outcome: Creatinine Clearance Following Administration of Oral Valacyclovir Suspension 20 mg/kg Every 8 Hours
Description: Blood will be collected to determine the drug concentration of acyclovir, the metabolite of valacyclovir and will include CL/F.
Time Frame: Between Day 2 and Day 7 of valacyclovir administration: 0, 1-2, 3-5 hours.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
L/h | 3.1 (1.8)

3. Primary Outcome: Half-life Following Administration of Oral Valacyclovir Suspension 20 mg/kg Every 8 Hours
Description: Blood will be collected to determine the drug concentration of acyclovir, the metabolite of valacyclovir and will include T1/2.
Time Frame: Between Day 2 and Day 7 of valacyclovir administration: 0, 1-2, 3-5 hours.
Measure: Mean (Standard Deviation); unit: hrs.
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
hrs. | 2.7 (1.2)

4. Secondary Outcome: Area Under the Curve Following Administration of Parenteral Acyclovir 20 mg/kg Every 8 Hours
Description: This study will determine the blood concentrations of acyclovir flowing valacyclovir administration. The goal is to define the valacyclovir dose which will allow a switch from IV to PO medication. In so doing, the potential duration of hospitalization can be decreased.
  To achieve this end, blood is collected to determine AUC.
Time Frame: One PK level drawn randomly on days 1-7; in addition, on one day between day 8 -14 of parenteral acyclovir, 3 PK levels to be drawn (drawn 30 minutes prior to infusion, 15 minutes after completion of infusion, and 3-4 hours after infusion)
Measure: Mean (Standard Deviation); unit: mgxh/L
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
mgxh/L | 70.1 (41)

5. Secondary Outcome: Half-life Following Administration of Parenteral Acyclovir 20 mg/kg Every 8 Hours
Description: This study will determine the blood concentrations of acyclovir flowing valacyclovir administration. The goal is to define the valacyclovir dose which will allow a switch from IV to PO medication. In so doing, the potential duration of hospitalization can be decreased.
  To achieve this end, blood is collected to determine T1/2 of drug.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
hrs | 2.5 (1.3)

6. Secondary Outcome: Creatinine Clearance Following Administration of Parenteral Acyclovir 20 mg/kg Every 8 Hours
Description: This study will determine the blood concentrations of acyclovir flowing valacyclovir administration. The goal is to define the valacyclovir dose which will allow a switch from IV to PO medication. In so doing, the potential duration of hospitalization can be decreased.
  To achieve this end, blood is collected to determine creatinine clearance of drug.
Time Frame: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
L/h | 1.1 (0.4)

7. Secondary Outcome: Comparison of the Area Under the Curve of 20 mg/kg IV Acyclovir to the Area Under the Curve of 20 mg/kg PO Valacyclovir
Description: To determine if the concentration of the active metabolite acyclovir after administration of acyclovir and valacyclovir at specified time intervals produces the same area under the curve
Time Frame: Random PK levels on days 1-7 of acyclovir administration, PK levels obtained on one day between day 8-14 at specified time intervals, and PK levels obtained one day while on valacyclovir (see outcome 1 and outcome 3 for time intervals)
Measure: Mean (Standard Deviation); unit: AUC- mgxh/l
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
Number analyzed (Participants) | 7
AUC- mgxh/l
  PO valacyclovir AUC | 28.8 (16.8)
  IV acyclovir AUC (linear adjustment) | 74 (41.0)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Neonatal HSV Disease Requiring Suppressive Therapy
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/92/NCT04448392/Prot_SAP_000.pdf